CLINICAL TRIAL: NCT02953314
Title: A Phase 3, Open Label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of VX-661 in Combination With Ivacaftor in Subjects 6 Through 11 Years of Age With Cystic Fibrosis, Homozygous or Heterozygous for the F508del CFTR Mutation
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of VX-661/Ivacaftor in Pediatric Subjects With Cystic Fibrosis (CF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX15-661-113; 2017-001164-38 (EudraCT Number)
Record Dates: First submitted 2016-10-18; First posted 2016-11-02 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): Participants weighing <25 kg received TEZ 50 mg once daily/IVA 75 mg q12h orally for 14 days.
  Participants weighing ≥25 kg received TEZ 50 mg once daily/IVA 150 mg q12h orally for 14 days.
  Interventions: Drug: TEZ; Drug: IVA
- Part B (Experimental): Participants weighing <40 kg received TEZ 50 mg/IVA 75 mg as fixed dose combination orally once daily in the morning and IVA 75 mg orally once daily in the evening for 24 weeks.
  Participants weighing ≥40 kg received TEZ 100 mg/IVA 150 mg as fixed dose combination orally once daily in the morning and IVA 150 mg orally once daily in the evening for 24 weeks.
  Interventions: Drug: TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: TEZ
  Other Names: tezacaftor; VX-661
  Arms: Part A
Drug: TEZ/IVA
  Other Names: tezacaftor/ivacaftor; VX-661/VX-770
  Arms: Part B
Drug: IVA
  Other Names: ivacaftor; VX-770

SUMMARY:
This is a Phase 3, 2-part (Part A and Part B), open label, multicenter study evaluating the pharmacokinetic (PK), safety, and tolerability of multiple doses of tezacaftor (TEZ) in combination with ivacaftor (IVA) in subjects 6 through 11 years of age with CF who are homozygous or heterozygous for the F508del- CF transmembrane conductance regulator protein (CFTR) mutation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who weigh ≥15 kg without shoes at the Screening Visit.
* All genotypes as specified by the study protocol are eligible in Part A.
* The following genotypes are eligible in Part B:

  * homozygous for the F508del CFTR mutation
  * heterozygous for the F508del CFTR mutation and with a second allele with a CFTR mutation predicted to have residual function.
  * heterozygous for the F508del CFTR mutation and with a second CFTR allele with a gating defect that is clinically demonstrated to be ivacaftor responsive
* Subjects with a confirmed diagnosis of CF defined as a sweat chloride value ≥60 mmol/L or chronic sinopulmonary and/or gastrointestinal disease consistent with a diagnosis of CF. Subjects who are homozygous for the F508del-CFTR mutation must have a sweat chloride value ≥60 mmol/L.
* Subjects with ppFEV1 of ≥40 percentage points at the Screening Visit
* Subjects with stable CF disease as deemed by the investigator at the Screening Visit.
* Subjects who are willing to remain on their stable CF medication regimen through Day 14 (Part A) or through Week 24 (Part B) or, if applicable, through the Safety Follow up Visit.
* Subjects who are able to swallow tablets.
* Female subjects of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Day 1 Visit before receiving the first dose of study drug.
* Subjects of childbearing potential who are sexually active must meet the contraception requirements

Exclusion Criteria:

* History of any comorbidity reviewed at the Screening Visit that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Any clinically significant laboratory abnormalities at the Screening Visit that would interfere with the study assessments or pose an undue risk for the subject.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 28 days before Day 1
* Colonization with organisms associated with a more rapid decline in pulmonary status.
* A standard 12 lead ECG demonstrating QTc >450 msec at the Screening Visit.
* History of solid organ or hematological transplantation at the Screening Visit.
* Ongoing or prior participation in an investigational drug study or use of commercially available CFTR modulator (except physician-prescribed Kalydeco for approved indications) within 30 days of screening.
* Use of restricted medication or food within a specified duration before the Screening Visit or first dose of study drug and/or unwillingness to maintain the restrictions.
* History or evidence of cataract, lens opacity, Y-suture, or lamellar rings determined to be clinically significant by the ophthalmologist during the ophthalmologic examination at the Screening Visit.
* Pregnant and nursing females.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (30):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Little Rock, Arkansas
  - Los Angeles, California
  - Palo Alto, California
  - Aurora, Colorado
  - Wilmington, Delaware
  - Orlando, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Manchester, New Hampshire
  - Buffalo, New York
  - New York, New York
  - Syracuse, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Walker S, Flume P, McNamara J, Solomon M, Chilvers M, Chmiel J, Harris RS, Haseltine E, Stiles D, Li C, Ahluwalia N, Zhou H, Owen CA, Sawicki G; VX15-661-113 Investigator Group. A phase 3 study of tezacaftor in combination with ivacaftor in children aged 6 through 11 years with cystic fibrosis. J Cyst Fibros. 2019 Sep;18(5):708-713. doi: 10.1016/j.jcf.2019.06.009. Epub 2019 Jun 26. PMID 31253540

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 2-parts (Part A and B). The planned primary analysis was designed to assess overall treatment arm "TEZ/IVA", irrespective of weight-based dosing regimen. The aim of weight based dosing is to achieve similar exposures in children of different weights, thus analysis is presented for the single treatment arm "TEZ/IVA".
Groups:
- Part A: Participants weighing <25 kg received TEZ 50 mg/IVA 75 mg for 14 days.
  Participants weighing ≥25 kg received TEZ 50 mg/IVA 150 mg for 14 days.
- Part B: Participants weighing <40 kg received TEZ 50 mg/IVA 75 mg as fixed dose combination in the morning and IVA 75 mg orally in the evening for 24 weeks.
  Participants weighing ≥40 kg received TEZ 100 mg/IVA 150 mg as fixed dose combination in the morning and IVA 150 mg in the evening for 24 weeks.
Period: Overall Study
Arm/Group | Part A | Part B
Started | 13 | 70
Completed | 13 | 67
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal of consent (not due to AE) | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Part B: Participants weighing <40 kg received TEZ 50 mg/IVA 75 mg as fixed dose combination in the morning and IVA 75 mg in the evening for 24 weeks.
  Participants weighing ≥40 kg received TEZ 100 mg/IVA 150 mg as fixed dose combination in the morning and IVA 150 mg in the evening for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 13 | 70 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 70 | 83
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 34 | 41
  Male | 6 | 36 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 13 | 67 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 68 | 80
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Maximum Observed Concentration (Cmax) of TEZ and IVA
Time Frame: Day 1 and Day 14
Population: Pharmacokinetic (PK) set included participants who received at least 1 dose of study drug and for whom the primary PK data were considered to be sufficient and interpretable. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A
Number analyzed (Participants) | 13
nanogram per milliliter (ng/mL)
  Day 1: TEZ (<25 Kg): number analyzed (Participants) | 2
  Day 1: TEZ (<25 Kg) | 6630 (10.3)
  Day 1: TEZ (≥25 Kg): number analyzed (Participants) | 11
  Day 1: TEZ (≥25 Kg) | 4310 (42.6)
  Day 14: TEZ (<25 Kg): number analyzed (Participants) | 2
  Day 14: TEZ (<25 Kg) | 6300 (10.3)
  Day 14: TEZ (≥25 Kg): number analyzed (Participants) | 10
  Day 14: TEZ (≥25 Kg) | 5340 (49.0)
  Day 1: IVA (<25 Kg): number analyzed (Participants) | 1
  Day 1: IVA (<25 Kg) | 656
  Day 1: IVA (≥25 Kg): number analyzed (Participants) | 9
  Day 1: IVA (≥25 Kg) | 1010 (64.3)
  Day 14: IVA (<25 Kg): number analyzed (Participants) | 2
  Day 14: IVA (<25 Kg) | 578 (60.4)
  Day 14: IVA (≥25 Kg): number analyzed (Participants) | 10
  Day 14: IVA (≥25 Kg) | 1490 (105)

2. Primary Outcome: Part A: Area Under the Concentration Versus Time Curve During Dosing Interval (AUCtau) of TEZ and IVA
Time Frame: Day 1 and Day 14
Population: PK set. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points."Number Analyzed=0" signified no subjects were evaluated for the specified parameter at that time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Part A
Number analyzed (Participants) | 13
hour*nanogram per milliliter (hr*ng/mL)
  Day 1: TEZ (<25 Kg): number analyzed (Participants) | 2
  Day 1: TEZ (<25 Kg) | 54300 (16.2)
  Day 1: TEZ (≥25 Kg): number analyzed (Participants) | 11
  Day 1: TEZ (≥25 Kg) | 41600 (36.2)
  Day 14: TEZ (<25 Kg): number analyzed (Participants) | 2
  Day 14: TEZ (<25 Kg) | 66500 (30.5)
  Day 14: TEZ (≥25 Kg): number analyzed (Participants) | 10
  Day 14: TEZ (≥25 Kg) | 71600 (61.1)
  Day 1: IVA (<25 Kg): number analyzed (Participants) | 0
  Day 1: IVA (≥25 Kg): number analyzed (Participants) | 0
  Day 14: IVA (<25 Kg): number analyzed (Participants) | 2
  Day 14: IVA (<25 Kg) | 5050 (49.1)
  Day 14: IVA (≥25 Kg): number analyzed (Participants) | 10
  Day 14: IVA (≥25 Kg) | 12400 (118)

3. Primary Outcome: Part B: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 28
Population: Safety set: included all participants who received at least 1 dose of study drug. The planned analysis was designed to assess overall treatment arm, irrespective of weight-based dosing regimen. The aim of weight based dosing is to achieve similar exposures in children of different weights, thus analysis is presented for the single treatment arm.
Measure: Number; unit: participants
Arm/Group | Part B
Number analyzed (Participants) | 70
participants
  Participants with AEs | 65
  Participants with SAEs | 6

4. Secondary Outcome: Part A: Cmax of TEZ Metabolites (M1-TEZ, M2-TEZ) and IVA Metabolites (M1-IVA, M6-IVA)
Time Frame: Day 1 and Day 14
Population: PK set. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A
Number analyzed (Participants) | 13
ng/mL
  Day 1: M1-TEZ (<25 kg): number analyzed (Participants) | 2
  Day 1: M1-TEZ (<25 kg) | 1720 (3.29)
  Day 1: M1-TEZ (≥25 kg): number analyzed (Participants) | 11
  Day 1: M1-TEZ (≥25 kg) | 1530 (22.0)
  Day 14: M1-TEZ (<25 kg): number analyzed (Participants) | 2
  Day 14: M1-TEZ (<25 kg) | 8360 (22)
  Day 14: M1-TEZ (≥25 kg): number analyzed (Participants) | 10
  Day 14: M1-TEZ (≥25 kg) | 5930 (19.9)
  Day 1: M2-TEZ (<25 kg): number analyzed (Participants) | 2
  Day 1: M2-TEZ (<25 kg) | 1130 (4.36)
  Day 1: M2-TEZ (≥25 kg): number analyzed (Participants) | 11
  Day 1: M2-TEZ (≥25 kg) | 922 (25.8)
  Day 14: M2-TEZ (<25 kg): number analyzed (Participants) | 2
  Day 14: M2-TEZ (<25 kg) | 6180 (27.2)
  Day 14: M2-TEZ (≥25 kg): number analyzed (Participants) | 10
  Day 14: M2-TEZ (≥25 kg) | 5350 (27.2)
  Day 1: M1-IVA (<25 kg): number analyzed (Participants) | 1
  Day 1: M1-IVA (<25 kg) | 2320
  Day 1: M1-IVA (≥25 kg): number analyzed (Participants) | 9
  Day 1: M1-IVA (≥25 kg) | 2430 (57.1)
  Day 14: M1-IVA (<25 kg): number analyzed (Participants) | 2
  Day 14: M1-IVA (<25 kg) | 1460 (34.6)
  Day 14: M1-IVA (≥25 kg): number analyzed (Participants) | 10
  Day 14: M1-IVA (≥25 kg) | 3420 (72.7)
  Day 1: M6-IVA (<25 kg): number analyzed (Participants) | 1
  Day 1: M6-IVA (<25 kg) | 849
  Day 1: M6-IVA (≥25 kg): number analyzed (Participants) | 9
  Day 1: M6-IVA (≥25 kg) | 1070 (55.7)
  Day 14: M6-IVA (<25 kg): number analyzed (Participants) | 2
  Day 14: M6-IVA (<25 kg) | 1090 (31.4)
  Day 14: M6-IVA (≥25 kg): number analyzed (Participants) | 10
  Day 14: M6-IVA (≥25 kg) | 2720 (59.2)

5. Secondary Outcome: Part A: AUCtau of TEZ Metabolites (M1-TEZ, M2-TEZ) and IVA Metabolites (M1-IVA, M6-IVA)
Time Frame: Day 1 and Day 14
Population: PK set. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points. "Number Analyzed=0" signified no subjects were evaluated for the specified parameter at that time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Part A
Number analyzed (Participants) | 13
hr*ng/mL
  Day 1: M1-TEZ (<25 kg): number analyzed (Participants) | 2
  Day 1: M1-TEZ (<25 kg) | 36500 (5.80)
  Day 1: M1-TEZ (≥25 kg): number analyzed (Participants) | 11
  Day 1: M1-TEZ (≥25 kg) | 27400 (26.3)
  Day 14: M1-TEZ (<25 kg): number analyzed (Participants) | 2
  Day 14: M1-TEZ (<25 kg) | 160000 (15.5)
  Day 14: M1-TEZ (≥25 kg): number analyzed (Participants) | 10
  Day 14: M1-TEZ (≥25 kg) | 121000 (17.1)
  Day 1: M2-TEZ (<25 kg): number analyzed (Participants) | 2
  Day 1: M2-TEZ (<25 kg) | 14200 (12.3)
  Day 1: M2-TEZ (≥25 kg): number analyzed (Participants) | 11
  Day 1: M2-TEZ (≥25 kg) | 11100 (25.9)
  Day 14: M2-TEZ (<25 kg): number analyzed (Participants) | 2
  Day 14: M2-TEZ (<25 kg) | 137000 (32.7)
  Day 14: M2-TEZ (≥25 kg): number analyzed (Participants) | 10
  Day 14: M2-TEZ (≥25 kg) | 119000 (27.7)
  Day 1: M1-IVA (<25 kg): number analyzed (Participants) | 0
  Day 1: M1-IVA (≥25 kg): number analyzed (Participants) | 0
  Day 14: M1-IVA (<25 kg): number analyzed (Participants) | 2
  Day 14: M1-IVA (<25 kg) | 13700 (52.1)
  Day 14: M1-IVA (≥25 kg): number analyzed (Participants) | 10
  Day 14: M1-IVA (≥25 kg) | 30300 (81.1)
  Day 1: M6-IVA (<25 kg): number analyzed (Participants) | 0
  Day 1: M6-IVA (≥25 kg): number analyzed (Participants) | 0
  Day 14: M6-IVA (<25 kg): number analyzed (Participants) | 2
  Day 14: M6-IVA (<25 kg) | 10200 (58.5)
  Day 14: M6-IVA (≥25 kg): number analyzed (Participants) | 10
  Day 14: M6-IVA (≥25 kg) | 26000 (70.6)

6. Secondary Outcome: Part A: Number of Participants With AEs and SAEs
Time Frame: Day 1 up to Day 28
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Part A
Number analyzed (Participants) | 13
participants
  Participants with AEs | 12
  Participants with SAEs | 0

7. Secondary Outcome: Part B: Cmax of TEZ, TEZ Metabolites (M1-TEZ, M2-TEZ), IVA, and IVA Metabolites (M1-IVA, M6-IVA)
Time Frame: Week 16
Population: PK set. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B
Number analyzed (Participants) | 69
ng/mL
  TEZ (<40 kg): number analyzed (Participants) | 62
  TEZ (<40 kg) | 4800 (33.7)
  TEZ (≥40 kg): number analyzed (Participants) | 7
  TEZ (≥40 kg) | 5870 (46.5)
  M1-TEZ (<40 kg): number analyzed (Participants) | 62
  M1-TEZ (<40 kg) | 5310 (36.0)
  M1-TEZ (≥40 kg): number analyzed (Participants) | 7
  M1-TEZ (≥40 kg) | 5440 (61.5)
  M2-TEZ (<40 kg): number analyzed (Participants) | 62
  M2-TEZ (<40 kg) | 4170 (47.4)
  M2-TEZ (≥40 kg): number analyzed (Participants) | 7
  M2-TEZ (≥40 kg) | 5210 (55.0)
  IVA (<40 kg): number analyzed (Participants) | 62
  IVA (<40 kg) | 725 (56.9)
  IVA (≥40 kg): number analyzed (Participants) | 7
  IVA (≥40 kg) | 886 (58.7)
  M1-IVA (<40 kg): number analyzed (Participants) | 62
  M1-IVA (<40 kg) | 1560 (54.8)
  M1-IVA (≥40 kg): number analyzed (Participants) | 7
  M1-IVA (≥40 kg) | 1870 (50.2)
  M6-IVA (<40 kg): number analyzed (Participants) | 62
  M6-IVA (<40 kg) | 870 (69.2)
  M6-IVA (≥40 kg): number analyzed (Participants) | 7
  M6-IVA (≥40 kg) | 1120 (29.5)

8. Secondary Outcome: Part B: AUCtau of TEZ, TEZ Metabolites (M1-TEZ, M2-TEZ), IVA, and IVA Metabolites (M1-IVA, M6-IVA )
Time Frame: Week 16
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Part B
Number analyzed (Participants) | 69
hr*ng/mL
  TEZ (<40 kg): number analyzed (Participants) | 61
  TEZ (<40 kg) | 50300 (36.3)
  TEZ (≥40 kg): number analyzed (Participants) | 6
  TEZ (≥40 kg) | 60900 (50.6)
  M1-TEZ (<40 kg): number analyzed (Participants) | 61
  M1-TEZ (<40 kg) | 104000 (44.2)
  M1-TEZ (≥40 kg): number analyzed (Participants) | 6
  M1-TEZ (≥40 kg) | 100000 (87.2)
  M2-TEZ (<40 kg): number analyzed (Participants) | 61
  M2-TEZ (<40 kg) | 88400 (57.0)
  M2-TEZ (≥40 kg): number analyzed (Participants) | 6
  M2-TEZ (≥40 kg) | 93600 (46.5)
  IVA (<40 kg): number analyzed (Participants) | 59
  IVA (<40 kg) | 5330 (62.2)
  IVA (≥40 kg): number analyzed (Participants) | 6
  IVA (≥40 kg) | 7410 (53.8)
  M1-IVA (<40 kg): number analyzed (Participants) | 59
  M1-IVA (<40 kg) | 12700 (55.9)
  M1-IVA (≥40 kg): number analyzed (Participants) | 6
  M1-IVA (≥40 kg) | 17200 (40.4)
  M6-IVA (<40 kg): number analyzed (Participants) | 59
  M6-IVA (<40 kg) | 8140 (70.2)
  M6-IVA (≥40 kg): number analyzed (Participants) | 6
  M6-IVA (≥40 kg) | 11100 (39.4)

9. Secondary Outcome: Part B: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Week 24
Population: FAS: participants who carry the intended CFTR mutations and received at least 1 dose of study drug. The aim of weight based dosing is to achieve similar exposures in children of different weights, thus the planned analysis is presented for the single treatment arm irrespective of weight-based dosing regimen.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Part B
Number analyzed (Participants) | 70
percentage points | 0.9 [-0.6 to 2.3]

10. Secondary Outcome: Part B: Relative Change in ppFEV1
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Part B
Number analyzed (Participants) | 70
percent change | 1.4 [-0.4 to 3.1]

11. Secondary Outcome: Part B: Absolute Change in Weight
Time Frame: From Baseline at Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Part B
Number analyzed (Participants) | 70
kg | 1.7 [1.3 to 2.0]

12. Secondary Outcome: Part B: Absolute Change in Weight-for-age Z-Score
Description: z-score is a statistical measure to describe whether a mean was above or below the standard. Weight, adjusted for age and sex, was analyzed as weight-for-age z-score. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher weight.
Time Frame: From Baseline at Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B
Number analyzed (Participants) | 70
z-score | 0.00 [-0.05 to 0.05]

13. Secondary Outcome: Part B: Absolute Change in Height
Time Frame: From Baseline at Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeter (cm)
Arm/Group | Part B
Number analyzed (Participants) | 70
centimeter (cm) | 2.7 [2.4 to 2.9]

14. Secondary Outcome: Part B: Absolute Change in Height-for-age z-Score
Description: z-score is a statistical measure to describe whether a mean was above or below the standard. Height, adjusted for age and sex, was analyzed as height-for-age z-score. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher height.
Time Frame: From Baseline at Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B
Number analyzed (Participants) | 70
z-score | 0.00 [-0.05 to 0.05]

15. Secondary Outcome: Part B: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kg divided by height in square meter (m^2).
Time Frame: From Baseline at Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Part B
Number analyzed (Participants) | 70
kg/m^2 | 0.23 [0.06 to 0.40]

16. Secondary Outcome: Part B: Absolute Change in BMI-for-age z-Score
Description: BMI was defined as weight in kg divided by height in m^2. z-score is a statistical measure to describe whether a mean was above or below the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher BMI.
Time Frame: From Baseline at Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B
Number analyzed (Participants) | 70
z-score | -0.03 [-0.10 to 0.04]

17. Secondary Outcome: Part B: Absolute Change in Sweat Chloride
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Week 4
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Part B
Number analyzed (Participants) | 70
millimole per liter (mmol/L) | -13.0 [-16.2 to -9.9]

18. Secondary Outcome: Part B: Absolute Change in Sweat Chloride
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Part B
Number analyzed (Participants) | 70
mmol/L | -14.5 [-17.4 to -11.6]

19. Secondary Outcome: Part B: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline through Week 24
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part B
Number analyzed (Participants) | 70
units on a scale | 3.4 [1.4 to 5.5]

ADVERSE EVENTS:
Time Frame: Part A: Day 1 up to Day 28; Part B: Day 1 up to Week 28
Description: Safety set: included all participants who received at least 1 dose of study drug. The planned analysis was designed to assess overall treatment arm, irrespective of weight-based dosing regimen. The aim of weight based dosing is to achieve similar exposures in children of different weights, thus analysis is presented for the single treatment arm for Part A and Part B.
Arm/Group | Part A | Part B
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/13 | 6/70
Other Adverse Events (participants affected / at risk) | 12/13 | 62/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=13) | Part B (N=70)
Constipation (Gastrointestinal disorders) | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=13) | Part B (N=70)
Abdominal pain (Gastrointestinal disorders) | 0 | 10
Abdominal pain upper (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 7
Constipation (Gastrointestinal disorders) | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 6
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 15
Influenza (Infections and infestations) | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 6
Acute sinusitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 5
Urinary tract infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 25
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Pyrexia (General disorders) | 1 | 13
Alanine aminotransferase increased (Investigations) | 0 | 6
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 3 | 6
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT02953314/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02953314/SAP_001.pdf